CLINICAL TRIAL: NCT03149588
Title: Comparison of Effects of Propofol and Sevoflurane as Maintaining Anesthetics During General Anesthesia on Maternal and Fetal Outcomes After Cesarean Section
Brief Title: Comparison of Propofol and Sevoflurane as Maintaining Anesthetics During General Anesthesia of Cesarean Section
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tao Zhang (Other)
Responsible Party: Sponsor-Investigator, Tao Zhang, Clinical Professor of Department of Anesthesiology, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GACS
Record Dates: First submitted 2017-05-05; First posted 2017-05-11 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Sevoflurane; Propofol; Cesarean Section
MeSH Terms: interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- propofol (Experimental)
  Interventions: Drug: propofol
- sevoflurane (Experimental)
  Interventions: Drug: sevoflurane

INTERVENTIONS:
Drug: propofol — Using propofol and remifentanil as maintenance of general anesthesia during caesarean section.
  Arms: propofol
Drug: sevoflurane — Using sevoflurane and remifentanil as maintenance of general anesthesia during caesarean section.
  Arms: sevoflurane

SUMMARY:
Sevoflurane and propofol are the most popular drug choices for maintenance of general anaesthesia for caesarean section. However, effects of these two anesthetics on maternal and fetal outcomes after caesarean section haven't been compared directly. The aim of this study is to compare the effects of sevoflurane and propofol as maintenance of general anesthesia, and to try to determine which anesthetic is better for maternal and fetal outcomes after caesarean section.

DETAILED DESCRIPTION:
General anaesthesia is mostly performed for emergency grade 1 caesarean section and due to a lack of time to apply a neuraxial anaesthesia technique. Rapid sequence induction using propofol and rocuronium should become the standard for general anaesthesia in the obstetric patient. Both sevoflurane and propofol are considered to be appropriate for the maintenance of general anaesthesia during caesarean section. However, effects of these two anesthetics on maternal and fetal outcomes after caesarean section haven't been compared directly in the past. And for most anaesthesiologists, the clinical experience with general anaesthesia for caesarean section is very low. This study is to compare the effects of sevoflurane and propofol as maintenance of general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASAⅠor Ⅱ parturients (aged 18-35 years) undergoing elective caesarean section

Exclusion Criteria:

* Parturients with severe pregnancy complications

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-04-03 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Maternal hospital stay | Before dismissed from hospital
  Maternal hospital stay time
Maternal mortality | Before dismissed from hospital
  Maternal mortality in hospital
Newborn hospital stay | Before dismissed from hospital
  Newborn hospital stay time
Newborn mortality | Before dismissed from hospital
  Newborn mortality in hospital

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital, Sun Yat-sen University, Guangzhou, China

REFERENCES:
- [Background] Devroe S, Van de Velde M, Rex S. General anesthesia for caesarean section. Curr Opin Anaesthesiol. 2015 Jun;28(3):240-6. doi: 10.1097/ACO.0000000000000185. PMID 25827280